CLINICAL TRIAL: NCT01520740
Title: Collateral Ventilation Effects on Response to AeriSeal System Treatment in Upper Lobe Predominant Emphysema
Acronym: CV+/-
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-C11-004PLV
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Pulmonary Emphysema
Keywords: Gold Stage III; Gold Stage IV; Chronic Obstructive Pulmonary Disease; COPD; Lung Volume Reduction Surgery; LVRS; Bronchoscopic Lung Volume Reduction; BLVR; Upper Lobe Predominant; ULP; Heterogeneous; Homogeneous
MeSH Terms: conditions — Pulmonary Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collateral Ventilation Positive (CV+) (Active Comparator)
  Interventions: Device: Emphysematous Lung Sealant
- Collateral Ventilation Negative (CV-) (Active Comparator)
  Interventions: Device: Emphysematous Lung Sealant

INTERVENTIONS:
Device: Emphysematous Lung Sealant — 4 Subsegments treated - 2 each bilaterally
  Other Names: AeriSeal System Treatment
  Arms: Collateral Ventilation Positive (CV+)
Device: Emphysematous Lung Sealant — 4 Subsegments treated - 2 each bilaterally
  Other Names: AeriSeal System Treatment
  Arms: Collateral Ventilation Negative (CV-)

SUMMARY:
This study will evaluate the effects of baseline collateral ventilation status on outcomes following treatment with AeriSeal System in patients with advanced upper-lobe predominant heterogenous emphysema.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent and to participate in the study
* Age > or = 40 years at the time of the screening
* Advanced upper lobe predominant emphysema by CT scan
* Two (2) subsegments appropriate for treatment based upon CT scan in 2 different upper lobe segments in each lung (total 4 available subsegments)
* MRCD questionnaire score of 2 or greater at screening
* Failure of medical therapy to provide relief of symptoms
* Spirometry 15 minutes after administration of bronchodilator (BOTH):

  * FEV1 < 50% predicted
  * FEV1/FVC ratio < 70%
* Lung volumes by plethysmography (BOTH):

  * TLC > 100% predicted
  * RV > 150% predicted
* DLco > or = 20 and < or = 60% predicted
* Oxygen saturation (SpO2) > 90% on < or = 4 L/min supplemental O2, at rest
* Six-Minute Walk Test distance > or = 150 m
* Abstinence from smoking for at least 16 weeks prior to screening

Exclusion Criteria:

* Prior lung volume reduction surgery, prior lobectomy or pneumonectomy, prior lung transplantation, prior airway stent placement, prior pleurodesis, or prior endobronchial lung volume reduction therapy of any type
* Requirement for ventilator support (invasive or non-invasive)
* Three (3) or more COPD exacerbations requiring hospitalization within 1 year of Screening visit or a COPD exacerbation requiring hospitalization within 8 weeks of Screening visit
* α-1 antitrypsin serum level of <80 mg/dl (immunodiffusion) or <11µmol/L (nephelometry) at Screening visit in the absence of enzyme replacement therapy. Patients with documented α-1 antitrypsin deficiency requiring replacement therapy are excluded from the study participation.
* Pulmonary hypertension, defined as:

  * Echocardiogram with estimated peak systolic pressure > 45 mmHg in the presence of tricuspid valve regurgitation stated in the echocardiogram report
  * If the echocardiogram shows peak systolic pressure > 45 mmHg, right heart catheterization is required to rule out pulmonary hypertension, defined as peak systolic pressure > 45 mmHg or mean pressure > 35 mmHg
* Clinically significant asthma (reversible airway obstruction) or bronchiectasis
* CT scan: Presence of the following radiologic abnormalities:

  * Pulmonary nodule on CT scan greater that 1.0 cm in diameter (Does not apply if present for 2 years or more without increase in size or if proven benign by biopsy/PET)
  * Radiologic picture consistent with active pulmonary infection, e.g., unexplained parenchymal infiltrate
  * Significant interstitial lung disease
  * Significant pleural disease
  * Giant bullous disease (a predominant bulla > 10 cm in diameter)
* Use of systemic steroids > 20 mg/day or equivalent, immunosuppressive agents, heparins, oral anticoagulants (e.g., warfarin, dicumarol; note: antiplatelet drugs including aspirin and clopidogrel are permitted) and investigational medications within 4 weeks of screening
* Allergy or sensitivity to medications required to safely undergo AeriSeal System treatment
* Participation in an investigational study of a drug, biologic, or device not currently approved for marketing within 30 days prior to the screening visit
* Body mass index < 15 kg/m2 or > 35 kg/m2
* Female patient pregnant or breast-feeding or planning to be pregnant in the next year
* Significant comorbidity that carries prohibitive risks or is associated with less than 2-year expected survival, including any of the following:

  * HIV/AIDS
  * Active malignancy
  * Stroke or TIA within 12 months of screening
  * Myocardial infarction within 12 months of screening
  * Congestive heart failure within 12 months of screening defined at clinical evidence of right or left hear failure or left ventricular ejection fraction < 45% on echocardiogram
* Any condition that the Investigator believes would interfere with the intent of the study or would make participation not in the best interest of the patient such as alcoholism, high risk for drug abuse or noncompliance in returning for follow-up visits

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in group mean post bronchodilator Forced Exhalation Volume in one second (FEV1) | 24 Weeks

SECONDARY OUTCOMES:
Change from Baseline in group mean 6 Minute Walk Test (6MWT) distance | 24 Weeks
Change from baseline in group mean health related quality of life | 24 Weeks
  Change from baseline in group mean health related quality of life, measured in terms of St. George's Respiratory Questionnaire (SGRQ) total domain score

CONTACTS AND LOCATIONS:
Overall Officials: Janine McDermott, MS CCRP, Study Director — Aeris Therapeutics
Locations (13):
- Germany (10):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Charite Campus Virchow-Klinikum, Berlin
  - Klinikum Coburg, Coburg
  - Klinikum Donaustauf, Donaustauf
  - Asklepios Fachkliniken Muenchen - Gauting, Gauting
  - Universitatsklinikum Halle, Halle
  - Asklepios Klinik Hamburg-Harburg, Hamburg
  - Thoraxklinik am Uniklinikum Heidelberg, Heidelberg
  - Sana Kliniken Luebeck, Lübeck
  - Medizinische Klinik und Poliklinik Grosshadern, München
- Israel (3):
  - Hadassah - Hebrew University Medical Center, Jerusalem
  - Carmel Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Tel Aviv